CLINICAL TRIAL: NCT02193646
Title: Endoscopic Size Assessment of Advanced Adenomatous Polyps; Inter Observer Variations
Brief Title: Endoscopic Size Assessment of Advanced Adenomatous Polyps
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ESA-2014
Record Dates: First submitted 2014-07-14; First posted 2014-07-17 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Adenoma Detection Rate Improvement in Screening Colonoscopy
Keywords: Colonoscopy; Adenoma; ADR; Screening Colon Cancer
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators are retrospectively comparing detection rates of adenomatous polyps, advanced adenomas, and size assessment of the polyps among Rush University Medical Center endoscopists. The investigators plan to review whether the size assessment of adenomatous polyps affected the surveillance protocols and if the location of polyps detected affected the detection rates.

DETAILED DESCRIPTION:
The study plans to compare detection rates of adenomatous as well as the sessile serrated polyps, advanced adenomas and size assessment of the polyps among the endoscopists at the study site. In addition, the study team aims to evaluate rates of advanced neoplasia on surveillance colonoscopy based on certain features on initial colonoscopy and patient characteristics, including specific high-risk histologic features and concurrent medication usage such as aspirin. In addition, patients with at least one adenoma on surveillance colonoscopy will be identified and regarded as cases. Cases will be compared against normal surveillance colonoscopy. The Controls will be selected on a 1:1 ratio. Aspirin use will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Presence of adenomatous polyps detected at endoscopy and diagnosed pathologically by tissue biopsy
* Have a colonoscopy at RUMC for screening purposes

Exclusion Criteria:

* Failure to meet inclusion criteria
* Previous diagnosis of IBD or colorectal cancer

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing screening colonoscopies at Rush University Medical Center.
Sampling Method: Probability Sample
Enrollment: 1930 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
Adenomatous Polyp Detection Rate | one year
  Assessing for advanced adenomas (including location).
Endoscopic Size Assessment Versus Pathological Size Assessment | one year
  Size of polyps at time of endoscopic procedure will be compared to the size of the same polyp by pathological assessment.

SECONDARY OUTCOMES:
Retroflexion as an indication of adenoma detection rate in colorectal cancer screening | one year
  Retroflexion is a common but not mandatory practice in colonoscopy which as not been systematically studied in terms of polyp detection. Charts will be reviewed to determine whether retroflexion was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Alsayid, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Amanda Lin, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Van J, Alsayid M, Ma K, Vemulapalli K, Rex D, Melson J. Impact of Cold Snare vs Cold Forceps Resection of Diminutive Adenomas on Segmental Incomplete Resection Rate. Am J Gastroenterol. 2023 Aug 1;118(8):1410-1418. doi: 10.14309/ajg.0000000000002289. Epub 2023 Apr 11. PMID 37040556
- [Result] Alsayid M, Van J, Ma K, Melson J. Segmental metachronous adenoma rate as a metric for monitoring incomplete resection in a colonoscopy screening program. Gastrointest Endosc. 2021 Aug;94(2):347-354. doi: 10.1016/j.gie.2021.01.046. Epub 2021 Feb 6. PMID 33561485
- See also: Segmental metachronous adenoma rate as a metric for monitoring incomplete resection in a colonoscopy screening program — https://pubmed.ncbi.nlm.nih.gov/33561485/
- See also: Impact of Cold Snare vs Cold Forceps Resection of Diminutive Adenomas on Segmental Incomplete Resection Rate — https://journals.lww.com/ajg/fulltext/2023/08000/impact_of_cold_snare_vs_cold_forceps_resection_of.23.aspx